CLINICAL TRIAL: NCT03382249
Title: Sonodynamic Therapy Manipulates Atherosclerosis Regression Trial on Patients With Carotid Atherosclerotic Plaques
Acronym: SMART-C
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: redesign
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Collaborators: Tsinghua University (Other)
Responsible Party: Principal Investigator, Ye Tian, Professor, MD, PhD, First Affiliated Hospital of Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ye Tian carotid
Record Dates: First submitted 2017-12-04; First posted 2017-12-22 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Carotid Atherosclerosis
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMC and pseudo-SDT (Placebo Comparator): Optimal medical care (OMC) and pseudo-SDT are administrated in this arm. OMC is established according to the standards established by the 2017 China Guidelines for the Diagnosis and Treatment of Carotid Artery Stenosis in order to promote best practices for risk factor management. Pseudo-SDT combines saline injection and obstructed ultrasound exposure on targeted lesions to simulate real SDT progression.
  Interventions: Combination Product: pseudo-SDT
- OMC and SDT (Experimental): OMC and sonodynamic therapy (SDT) are administrated in this arm.
  Interventions: Combination Product: Sonodynamic therapy (SDT)

INTERVENTIONS:
Combination Product: Sonodynamic therapy (SDT) — Sonodynamic therapy(SDT) treatment is the combination of sonosensitizer administration and target atherosclerotic lesions ultrasound exposure. Sinoporphyrin sodium (DVDMS) as sonosensitizer, is dissolved in 0.9% sodium solution for following skin test and intravenous injection. 0.01mg/ml DVDMS solution (0.1ml) is prepared for skin test followed by 0.04 mg/ml DVDMS solution intravenous injection (0.2mg/kg).The target atherosclerotic lesions are marked on the corresponding skin with ultrasound guidance and underwent ultrasound exposure after 4 hours incubation. The therapeutic ultrasonic transducer is fixed to the marked skin site for 15min of each lesion. Ultrasound parameters included intensity of 1.6W/cm2 for carotid lesions, resonance frequency: 1.0 MHz and duty factor: 30%.
  Arms: OMC and SDT
Combination Product: pseudo-SDT — Pseudo-SDT combines saline injection and obstructed ultrasound exposure on targeted lesions to simulate real SDT progression.
  Arms: OMC and pseudo-SDT

SUMMARY:
Sonodynamic therapy (SDT) is a new treatment for carotid atherosclerotic plaque. The aim of this study is to assess the safety and efficacy of this technique.

DETAILED DESCRIPTION:
Carotid atherosclerotic plaque is an important cause of ischemic stroke, causes about 30% stroke/TIA attacks. Patients with carotid stenosis face an escalated risk of MI, PAD, and death. Treatments for patients with carotid plaque include lifestyle changes, medical management(such as control of hyperlipidemia, hypertension, and diabetes) and carotid revascularization(carotid endarterectomy or carotid artery stenting). Studies have suggested that plaque morphology and composition are important determinants of plaque stability, using serial MR imaging of the carotid artery allowed observation of changes in plaque composition. Contrast enhanced ultrasound (CEUS) is a well accepted technique for detection of intraplaque neovascularization(IPN) in carotid atherosclerotic disease.

The aim of this trial is to assess the safety and efficacy of SDT. The SDT can induce macrophage elimination and inhibiting matrix degradation, which will promote plaque lipid depletion, inflammation level decrease and changes in other plaque tissue components, leading to plaque stabilization and reduction.

An estimated 80 eligible patients will be randomly divided into two groups: optimal medical care (OMC) combined with pseudo-SDT and OMC combined with SDT. Recruitment will be performed over 1 year and patients will be followed for 3 months; the anticipated total study duration will be 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 80 years
* Carotid artery with 30%~70% stenosis by ultrasound and plaque thickness>2.5mm
* Patients without transient ischemic attack, minor stroke or amaurosis fugax within 6 months
* Patients' LDL-c level below 100 mg/dL(2.6mmol/L), well-controlled blood pressure(systolic BP<140 and diastolic BP<90 under resting conditions) and diabetes(HbA1c<7%)
* Written informed consent

Exclusion Criteria:

* Non-atherosclerotic carotid artery stenosis
* Contraindication to MRI( uses pacemaker, has metallic implants, claustrophobia)
* Acute MI, acute coronary syndrome or stroke within 4 weeks prior to visit or during run-in
* Severe cerebral artery stenosis, atrial fibrillation or MRI detected thrombosis that would cause stroke
* Previous significant adverse reaction to a statin
* Systemic disorders such as hepatic, renal, hematologic, and malignant disease
* Medical history that might limit the individual's ability to take trial treatments for the duration of the study
* Allergic to DVDMS or sonovue
* Diagnosis of porphyria
* Pregnant women and nursing mothers
* History of bilateral carotid endarterectomy or has immediate plans for carotid endarterectomy
* Not willing to be randomized into the 3 months trial
* Patient who is attending other clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Change in plaque LRNC volume, as assessed by MRI | Measured at Baseline, 1, 3 months
  The changes in plaque lipid-rich necrotic core (LRNC) volume as assessed by MRI.

SECONDARY OUTCOMES:
Change in plaque FT volume, as assessed by MRI | Measured at Baseline, 1, 3 months
  The changes in plaque fibrous tissue(FT) volume as assessed by MRI.
Change in IPH volume, as assessed by MRI | Measured at Baseline, 1, 3 months
  The changes in intraplaque hemorrhage (IPH) volume as assessed by MRI.
Change in calcification volume, as assessed by MRI | Measured at Baseline, 1, 3 months
  The changes in calcification volume as assessed by MRI.
Change in the status of fibrous cap, as assessed by MRI | Measured at Baseline, 1, 3 months
  The status of fibrous cap can be differentiated as thin/thick/ruptured assessed by MRI.
Change in plaque burden, as assessed by MRI | Measured at Baseline, 1, 3 months
  The plaque burden including wall volume(mm3), vessel wall thicknesses(VWT)(mm) and percent wall volume(PWV)(%) .
Change in MVE, as assessed by CEUS | Measured at Baseline, 1, 3 months
  The changes in normalised maximal video-intensity enhancement (MVE) are calculated to quantify the density of IPN as assessed by CEUS.
Change in peak flow velocity, as assessed by doppler ultrasound | Measured at Baseline, 1, 3 months
  The changes of the systolic and diastolic peak flow velocity of the affected segments by doppler ultrasound.
MACCE | Measured at Baseline, 1, 3 months
  incidence of major adverse cardiovascular and cerebrovascular events(MACCE)
Incidence of adverse events | Measured at Baseline, 1, 3 months
  Allergic to sunshine,hepatic or renal dysfunction,thyroid dysfunction
Lipid change | Measured at Baseline, 1, 3 months
  To evaluate the change in lipid and lipoprotein levels as assessed by percentage change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: TIAN YE, Study Chair — First Affiliated Hospital of Harbin Medical University
Locations (1):
- The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China